CLINICAL TRIAL: NCT02727504
Title: Low Flow Low Gradient Aortic Stenosis Relevance of the (re)Search for a Contractile Reserve
Acronym: LOWAS
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-A00896-43; 35RC15_9884_LOWAS (Other: CHU de Rennes)
Record Dates: First submitted 2016-03-21; First posted 2016-04-04 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic valve stenosis; low flow; dobutamine stress echocardiography
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Electrocardiography; Echocardiography, Three-Dimensional; Echocardiography, Stress; Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patient with aortic valve stenosis: 115 patients will undergo a medical examination in order to analyse their medical history, cardiovascular parameters and check inclusion and non-inclusion criterions.
  Then will be performed :
  * An electrocardiogram
  * 2D and 3D echocardiography
  * Dobutamine stress echocardiography
  * Blood tests : blood electrolytes, creatinine, hemoglobin, N-terminal pro-brain natriuretic peptide (NT-ProBNP), C reactive protein (CRP), soluble suppression of tumorigenicity-2 (ST-2)
  * A cardiac MRI
  * A cardiac scanner
  * A 6-minutes walking test
  * An evolution of the Duke Activity Score
  Interventions: Device: Electrocardiogram; Device: 2D and 3D echocardiography; Device: Dobutamine stress echocardiography; Biological: Blood tests; Device: Cardiac MRI; Device: Cardiac scanner; Other: 6-minutes walking test; Other: Duke Activity Score

INTERVENTIONS:
Device: Electrocardiogram — ECG at inclusion and M12
Device: 2D and 3D echocardiography — 2D and 3D echocardiography at inclusion and M12
Device: Dobutamine stress echocardiography — dobutamine stress echocardiography at inclusion
Biological: Blood tests — Blood test electrolytes, creatinine, hemoglobin, NT-proBNP, CRP, ST-2 at inclusion and M12
Device: Cardiac MRI — Cardiac MRI at inclusion
Device: Cardiac scanner — Cardiac scanner at inclusion
Other: 6-minutes walking test — 6-minutes walking test at inclusion and M12
Other: Duke Activity Score — Duke Activity Score at inclusion and M12

SUMMARY:
Investigators sought to demonstrate that the increase in the stroke volume during a dobutamine stress echocardiography might impact the prognosis of a patient addressed for a low flow low gradient suspected severe aortic valve stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient from 45 to 90 years old
* Patient agreeing freely to participate in the study
* Aortic surface area suspected to be < 1 cm² or < 0.6 cms²/m²
* Low aortic gradient defined by a mean pressure gradient < 40 mmHg
* Aortic low flow defined by: a stroke volume indexed < 35 ml/m2
* Any contra-indication for the realization of the MRI

Exclusion Criteria:

* Heart rhythm disorders
* Presence of comorbidity altering the 2-year prognosis of a patient (cancer, terminal renal insufficiency (GFR 30 ml / min / 1,73m2), liver cirrhosis, respiratory insufficiency (VEMS 1 L)
* Presence of a concomitant valvular heart disease with stenosis or regurgitation > moderated
* Persons subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with low flow low gradient aortic stenosis
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2016-05-11; Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Number of death of all cause | Month 12
Number of emergent hospitalization for any cardiovascular reason | Month 12

SECONDARY OUTCOMES:
Death (all causes) | 12 months
Emergency Cardiovascular hospitalization | 12 months
Change in left ventricular ejection fraction (LVEF), in global longitudinal strain in 2D and or 3D echocardiography | Inclusion, 12 months
Symptoms evolution | Inclusion, 12 months
  6-minute walking test
Symptoms evolution | Inclusion, 12 months
  Duke Activity Score

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No